CLINICAL TRIAL: NCT02167269
Title: Comparison of Minimal Fresh Gas Requirements of Baby EAR and Jackson Rees Anesthetic Circuit for General Anesthesia in Spontaneously Breathing Children Undergoing Surgery
Brief Title: Comparison of Minimal Fresh Gas Requirements of Baby EAR and Jackson Rees Anesthetic Circuit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Thepakorn Sathitkarnmanee, Associate professor, Khon Kaen University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HE531147
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Anesthesia
Keywords: enclosed afferent reservoir; Jackson Rees system; anesthesia breathing circuit; spontaneous breathing; pediatric anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baby EAR-JR (Active Comparator): The subjects receive Baby EAR circuit from the start until primary and secondary outcomes are achieved. Then the fresh gas flow will be increased to 500 ml/kg/min for 10 minutes before switching to Jackson-Rees (JR) circuit and the procedure will be repeated.
  Interventions: Device: Baby EAR
- JR-Baby EAR (Active Comparator): The subjects receive Jackson-Rees (JR) circuit from the start until primary and secondary outcomes are achieved. Then the fresh gas flow will be increased to 500 ml/kg/min for 10 minutes before switching to Baby EAR circuit and the procedure will be repeated.
  Interventions: Device: Baby EAR

INTERVENTIONS:
Device: Baby EAR — A modification of the Enclosed Afferent Reservoir anesthesia circuit (EAR) for pediatric use by adding a KKU one-way valve in the expiratory limb

SUMMARY:
The investigators invented the baby enclosed afferent reservoir anesthesia circuit (Baby EAR) which could be used safely in children between 5 and 20 kg, using a fresh gas flow of 2.5 and 3 L/min in the spontaneous breathing and controlled breathing, respectively. There has as yet been no study comparing the minimal fresh gas flow between the Baby EAR and Jackson-Rees anesthesia circuit (JR).

DETAILED DESCRIPTION:
After intubation, a caudal block with 0.25% bupivacaine with adrenaline :200,000 0.5 to 1 mL/kg was done. Anesthesia was maintained with a 50% N2O/O2 combination with sevoflurane 1 to 3%, adjusted to ensure a proper anesthetic level to achieve normal vital signs and to keep the end-tidal CO2 (ETCO2) <60 mmHg. Fentanyl 1 μg/kg/h was infused during the procedure. All patients were pontaneously ventilated with FGF 500 mL/kg/min at the start of each anesthesia breathing circuit, waiting for the depth of anesthesia to be maintained and the patient to spontaneously breathe for at least 10 minutes. Baseline ETCO2 and imCO2 were then measured. The pulse rate, blood pressure and respiratory rate were recorded every five minutes.

The FGF was reduced by 50 mL/kg/min every five minutes, waiting for the imCO2 to be regularly maintained at least 60 sec. The ETCO2 and imCO2 values were recorded until rebreathing occurred (imCO2 >2 mmHg) and measurements continued until rebreathing was not clinically acceptable (imCO2 >6 mmHg). The minimal FGF before rebreathing occurred (FGF of imCO2 ≤2 mmHg) is the amount of gas that does not cause rebreathing. The minimal FGF for which rebreathing was still acceptable (FGF of imCO2 ≤6 mmHg) is the amount of gas that was clinically acceptable. After switching the anesthesia breathing circuit, the FGF was increased to 500 mL/kg/min for 10 minutes and the procedure was repeated. The minimal FGF before the rebreathing occurred and the FGF at hich rebreathing was still clinically acceptable were recorded. After extubation, all of the patients were observed in the PACU and relevant factors recorded until there was good recovery from anesthesia before sending the patient back to the ward.

ELIGIBILITY:
Inclusion Criteria:

* weight between 5 and 20 kg
* ASA physical status I or II
* scheduled for general anesthesia

Exclusion Criteria:

* has respiratory or cardiovascular disease
* can not breathe spontaneously during anesthesia
* for whom the caudal block can not be done

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
inspired minimum CO2 (imCO2) > 2 mmHg | 2 hours
  All patients were spontaneously ventilated with FGF 500 ml/kg/min at the start of each anesthesia breathing circuit then reduced by 50 ml/kg/min every 5 min, waiting for the imCO2 to be regularly maintained at least 60 sec. The imCO2 values were recorded until rebreathing occurred (imCO2 > 2 mmHg)

SECONDARY OUTCOMES:
inspired minimum CO2 (imCO2) > 6 mmHg | 2 hours
  All patients were spontaneously ventilated with FGF 500 ml/kg/min at the start of each anesthesia breathing circuit reduced by 50 ml/kg/min every 5 min, waiting for the imCO2 to be regularly maintained at least 60 sec. The imCO2 values were recorded until rebreathing was not clinically acceptable (imCO2 > 6 mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: Sanchai Theerapongpakdee, MD, Principal Investigator — Faculty of Medicine, Khon Kaen University
Locations (1):
- Srinagarind Hospital, Khon Kaen, Thailand